CLINICAL TRIAL: NCT05629390
Title: Randomized Controlled, Multicenter, Double-Masked, Parallel Phase III Trial to Evaluate the Efficacy and Safety of Lotilaner Ophthalmic Solution for the Treatment of Demodex Blepharitis in China With an Open-Label Pharmacokinetics Sub-Study
Brief Title: Trial to Evaluate the Efficacy and Safety of TP-03, LIBRA Study
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: LianBio LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LB4001-301
Record Dates: First submitted 2022-11-17; First posted 2022-11-29 (Actual); Last update posted 2024-05-21 (Actual); Status verified 2024-05

CONDITIONS: Blepharitis
Keywords: Blepharitis
MeSH Terms: conditions — Blepharitis | interventions — lotilaner

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lotilaner Ophthalmic Solution (TP-03) (Experimental): Lotilaner Ophthalmic Solution (TP-03)
  Interventions: Drug: Lotilaner
- Vehicle Control (Placebo Comparator): Vehicle Control
  Interventions: Drug: Vehicle Control

INTERVENTIONS:
Drug: Lotilaner — Lotilaner Ophthalmic Solution
  Other Names: TP-03; S-Misoxam
  Arms: Lotilaner Ophthalmic Solution (TP-03)
Drug: Vehicle Control — Vehicle of TP-03 ophthalmic solution
  Arms: Vehicle Control

SUMMARY:
The Phase III main study is a randomized, controlled, multicenter, double blind, trial to evaluate the efficacy and safety of TP-03 (lotilaner ophthalmic solution, 0.25%), for the treatment of Demodex blepharitis in Chinese patients. The PK sub-study is a single-arm, open-label trial to evaluate systemic TP-03 in whole blood following topical ocular administration

DETAILED DESCRIPTION:
The main study is designed to demonstrate the superiority of TP-03 compared to vehicle for the treatment of Demodex blepharitis in Chinese patients. The vehicle of TP-03 was selected as the control since there are no approved pharmaceutical treatments for Demodex blepharitis. The vehicle as the control will provide evidence that the active ingredient is responsible for the response, not the vehicle alone.

A pharmacokinetics (PK) sub-study is included in the overall study design to evaluate systemic PK parameters of TP-03 in Chinese participants with Demodex blepharitis. The PK sub-study sites are separate from those of the Phase III study as described above.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, aged ≥ 18 years of age.
2. Be willing to sign the informed consent and deemed capable of complying with the requirements of the study protocol.
3. Has blepharitis
4. Stated willingness to comply with all study procedures and availability for the duration of the study.

Exclusion Criteria:

1. Have used lid hygiene products (e.g., lid scrubs) within 14 days of Screening or unwilling to forego the use of lid hygiene products during the study.
2. Have initiated treatment with an ocular topical prostaglandin analogue within 30 days of Screening or have any plans to change or discontinue treatment during the study
3. Pregnancy or lactation.
4. Any intraocular surgery (including ocular surface surgery, cataract surgery and intravitreal injection) or periocular surgery within 60 days prior to randomization, or any planned ocular surgical procedure during the study period
5. Have any unstable or uncontrolled, cardiac, pulmonary, renal, oncological, neurological, metabolic or other systemic condition that, in the opinion of the investigator, would possibly require the participant to seek emergent medical treatment during the course of this study. This includes, but is not limited to, unstable or uncontrolled cardiac arrhythmias, hypertension, coagulopathies, renal failure or advanced diabetes mellitus.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 163 (Actual)
Dates: Start 2022-10-23 (Actual); Primary Completion 2023-09-15 (Actual); Study Completion 2024-04-02 (Actual)

PRIMARY OUTCOMES:
The proportion of participants cured based on their collarette score of 0 for the upper eyelid of the analysis eye. | 43 days
  To demonstrate the efficacy of 0.25% Lotilaner Ophthalmic Solution to eliminate collarettes and eradicate mite in Demodex blepharitis
The proportion of participants with Demodex eradication based on the mite density of 0 mites/lash for the analysis eye at Day 43 | 43 days
  To demonstrate the efficacy of 0.25% Lotilaner Ophthalmic Solution to eliminate collarettes and eradicate mite in Demodex blepharitis
The assessment of treatment-related adverse effects | 43 days
  To demonstrate the safety of 0.25% TP-03 in Demodex blepharitis

SECONDARY OUTCOMES:
The proportion of participants cured based on a composite of collarette score of 0 and erythema score of 0 for the upper eyelid of the analysis eye | 43 days
  To demonstrate the efficacy of TP-03 to eliminate collarettes and erythema from the eyelid margin
Blood drug concentration of Lotilaner at Day 43 | 43 days
  To evaluate the blood drug concentration of Lotilaner following topical ocular administration of TP-03administration of 0.25% TP-03

CONTACTS AND LOCATIONS:
Overall Officials: Zuguo Liu, M.D, Principal Investigator — Xiamen Eye Center of Xiamen University
Locations (21):
- China (21):
  - Beijing Tongren Hospital, Beijing, Beijing Municipality
  - Peking University Third Hospital, Beijing, Beijing Municipality
  - Chongqing Aier Eye Hospital, Chongqing, Chongqing Municipality
  - Xiamen Eye Center of Xiamen University, Xiamen, Fujian
  - Guangzhou Aier Eye Hospital, Guangzhou, Guangdong
  - Zhongshan Ophthalmic Center, Sun Yat-sen University, Guangzhou, Guangdong
  - Hainan Eye Hospital, Haikou, Hainan
  - The First Affiliated Hospital of Harbin Medical University, Harbin, Heilongjiang
  - Henan Provincial Eye Hospital, Zhengzhou, Henan
  - Union Hospital, Tongji Medical College Huazhong University of Science and Technology, Wuhan, Hubei
  - Renmin Hospital of Wuhan University, Wuhan, Hubei
  - The Second Xiangya Hospital of Central South University, Changsha, Hunan
  - Xiangya Hospital, Central South University, Changsha, Hunan
  - The First Affiliated Hospital of University of South China, Hengyang, Hunan
  - Wuxi Second People's Hospital, Wuxi, Jiangsu
  - Eye& Ent Hospital of Fudan University, Shanghai, Shanghai Municipality
  - Shanghai General Hospital, Shanghai, Shanghai Municipality
  - Shanxi Provincial Eye Hospital, Taiyuan, Shanxi
  - Tianjin Medical University Eye Hospital, Tianjin, Tianjin Municipality
  - The Second Affiliated Hospital Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - Eye Hospital, Wenzhou Medical University, Wenzhou, Zhejiang